CLINICAL TRIAL: NCT07239492
Title: Efficacy and Safety Evaluation of Transcranial Non-invasive Temporal Interference Stimulation for Blood Pressure Regulation: A Pilot, Prospective Study
Brief Title: Efficacy and Safety Evaluation of Non-invasive Temporal Interference Stimulation for Blood Pressure Regulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liankun_Ren, Professor, Xuanwu Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-220-002
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Hypertension; Hypotension
Keywords: hypertension; temporal in terference; hypotension
MeSH Terms: conditions — Hypertension; Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temporal interference stimulation (Experimental): Patients with hypertension/hypotension assigned to temporal interference stimulation for 20 min per session.
  Interventions: Other: Temporal Interference

INTERVENTIONS:
Other: Temporal Interference — The intervention will consist of 5 days of 20-min temporal interference stimulation.

SUMMARY:
The primary objective of this research is to study the efficacy and safety of temporal interference stimulation for regulating the blood pressure.

DETAILED DESCRIPTION:
This project aims to include 25 participants, and evaluate the effectiveness and safety of temporal interference stimulation in patients with hypertension and hypotension through A pilot, prospective clinical trial. It is expected to provide new therapeutic options for patients with hypertension and hypotension with alternative treatment options.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 years old, male or female;
2. Three groups of patients will be enrolled in the study:

   1. Essential Hypertension Grade 1 (Low Risk) - Antihypertensive Medication-Naive Group: No other cardiovascular risk factors or disease history, with systolic blood pressure (SBP) ≥140 mmHg and <160 mmHg and/or diastolic blood pressure (DBP) ≥90 mmHg and <100 mmHg;
   2. Essential Hypertension - Refractory Hypertension Group: Meeting one of the following conditions after intensive lifestyle intervention plus taking 3 different types of antihypertensive drugs (including thiazide diuretics) for ≥4 weeks, with each drug at the maximum dose or maximum tolerated dose: Clinic blood pressure ≥140/90 mmHg and 24-hour average ambulatory blood pressure ≥130/80 mmHg, or average home blood pressure ≥135/85 mmHg; or blood pressure can only be controlled below 140/90 mmHg with ≥4 types of antihypertensive drugs;
   3. Neurogenic Orthostatic Hypotension (nOH) Group: A decrease in SBP ≥20 mmHg and/or DBP ≥10 mmHg within 3 minutes of the head-up tilt test (HUTT) and/or standing activity;
3. BMI: 18-30;
4. After being informed of the potential risks, the patient agrees to participate in this study and signs the informed consent form (ICF).

Exclusion Criteria:

1. Patients with secondary hypertension;
2. Patients with intracranial structural lesions (e.g., infarcts, vascular malformations, space-occupying lesions, etc.);
3. Pregnant women;
4. Individuals unable to cooperate due to mental illness or other reasons;
5. Those who have participated in other clinical studies within the past 3 months;
6. Patients who apply to withdraw from this clinical study for any reason;
7. Patients with cardiac insufficiency;
8. Patients excluding those with white coat effect;
9. Individuals with a high risk of cerebrovascular disease confirmed by transcranial magnetic resonance imaging (MRI).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure (BP24) | Up to 12 weeks after temporal interference stimulation
  Blood Pressure (BP24) is defined as 24-hour ambulatory blood pressure monitoring in each 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Liankun Ren, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital,Capital Medical University, Beijing, Beijing 100053, Beijing, China

IPD SHARING:
Plan to Share IPD: No